CLINICAL TRIAL: NCT01360567
Title: Taipei City Hospital, Taipei, Taiwan
Brief Title: The Effect of Green Tea Extract on Type 2 Diabetes With Hyperlipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taipei City Hospital (Other Government)
Collaborators: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Chung-Hua Hsu, chief medical officer, Taipei City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100002-63-020; TCH-971103 (Other Grant/Funding Number: CCMP100-RD-014); TCHIRB-971103 (Other Grant/Funding Number: CCMP100-RD-014)
Record Dates: First submitted 2011-05-20; First posted 2011-05-25 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Type 2 Diabetes; Hyperlipidemia
Keywords: green tea; EGCG; type 2 diabetes; hyperlipidemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperlipidemias | interventions — Tea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B formula (Placebo Comparator): placebo
  Interventions: Dietary Supplement: Placebo
- A formula (Experimental): Green tea extract
  Interventions: Dietary Supplement: Green tea extract

INTERVENTIONS:
Dietary Supplement: Green tea extract — 500 mg . one capsule of green tea extract, 3 times per day
  Other Names: EGCG: Green tea extract
  Arms: A formula
Dietary Supplement: Placebo — 500 mg . one capsule of placebo, 3 times per day
  Arms: B formula

SUMMARY:
The aim of the study is to examine whether the extract of green tea is effective on type 2 diabetes and hyperlipidemia.

DETAILED DESCRIPTION:
Percent change Homa insulin resistance, cholesterol and triglycerol.

ELIGIBILITY:
Inclusion Criteria:

* Age 20--69 years old
* Type 2 diabetes for > one year
* TG >= 150 mg/dl or LDL >= 100 mg/dl

Exclusion Criteria:

* GPT > 80 mg/dl
* Creatinine > 1.8 mg/dl
* Pregnancy
* AMI
* Stroke
* Operational or any not suitable patients diagnosis physician in charge

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Percent change of HOMA insulin resistance and TG | 16 weeks

SECONDARY OUTCOMES:
Percent change of HbA1C and Cholesterol | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Hua Hsu, MD, PhD, Principal Investigator — Taipei City Hospital
Locations (2):
- Taiwan (2):
  - Chung-Hua Hsu, Taipei
  - Taipei City Hospital, Taipei

REFERENCES:
- [Background] Hsu CH, Tsai TH, Kao YH, Hwang KC, Tseng TY, Chou P. Effect of green tea extract on obese women: a randomized, double-blind, placebo-controlled clinical trial. Clin Nutr. 2008 Jun;27(3):363-70. doi: 10.1016/j.clnu.2008.03.007. Epub 2008 May 12. PMID 18468736
- [Derived] Liu CY, Huang CJ, Huang LH, Chen IJ, Chiu JP, Hsu CH. Effects of green tea extract on insulin resistance and glucagon-like peptide 1 in patients with type 2 diabetes and lipid abnormalities: a randomized, double-blinded, and placebo-controlled trial. PLoS One. 2014 Mar 10;9(3):e91163. doi: 10.1371/journal.pone.0091163. eCollection 2014. PMID 24614112